CLINICAL TRIAL: NCT00475540
Title: A Randomized Clinical Trial of Vaginal Mesh for Prolapse
Brief Title: Efficacy Study of Vaginal Mesh for Prolapse
Acronym: VAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-232
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-07

CONDITIONS: Pelvic Organ Prolapse; Uterine Prolapse; Vaginal Prolapse; Cystocele; Rectocele
Keywords: prolapse; uterus; pelvic organ; vaginal prolpase
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse; Cystocele; Rectocele; Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolift mesh (Active Comparator): vaginal prolapse repair with mesh
  Interventions: Device: synthetic monofilament polypropylene mesh
- Prolapse repair without mesh (Active Comparator): vaginal prolapse repair without mesh
  Interventions: Device: synthetic monofilament polypropylene mesh

INTERVENTIONS:
Device: synthetic monofilament polypropylene mesh — Vaginal prolapse repair with mesh
  Other Names: Prolift

SUMMARY:
The primary aim of this double-blind, randomized clinical trial (RCT) is to test the hypothesis that the addition of a standardized technique of interpositional synthetic polypropylene mesh placement improves the one-year outcome of vaginal reconstructive surgery for pelvic organ prolapse compared to traditional vaginal reconstructive surgery without mesh.

DETAILED DESCRIPTION:
Minimally invasive surgical procedures using mesh have rapidly developed in the field of pelvic floor reconstruction. Unfortunately, safety and efficacy data have lagged behind the technical advancements. No randomized controlled trials of different vaginal apical suspension procedures have been reported. The use of synthetic vaginal mesh has evolved due to the 20-30% recurrence rate for conventional pelvic reconstructive surgeries. This trial will examine synthetic monofilament polypropylene mesh use in vaginal reconstructive surgery for vaginal Stage II-IV prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Woman > 21 yrs
* Stage II-IV vaginal prolapse
* Desires vaginal reconstructive surgery
* Able to complete study questionnaires and assessments
* Uterus < 12 weeks size
* Available for 12 months follow-up

Exclusion Criteria:

* Medical contraindications, e.g. current urinary tract, vaginal or pelvic infection, history of pelvic irradiation, history of lower urinary tract malignancy, chronic steroid use or a compromised immune system.
* Current intermittent catheterization.
* Pregnancy or desire for future fertility.
* Presence of an adnexal mass.
* Shortened vagina or other known Mullerian anomaly (e.g. uterine didelphys).
* Other laparoscopic or abdominal/pelvic surgery in the past 3 months.
* Known neurologic or medical condition affecting bladder function, e.g. Multiple Sclerosis, spinal cord injury.
* Need for concomitant surgery requiring an abdominal incision.
* < 12 months post-partum.
* Non-english speaking

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Iglesia, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Gutman RE, Nosti PA, Sokol AI, Sokol ER, Peterson JL, Wang H, Iglesia CB. Three-year outcomes of vaginal mesh for prolapse: a randomized controlled trial. Obstet Gynecol. 2013 Oct;122(4):770-777. doi: 10.1097/AOG.0b013e3182a49dac. PMID 24084533
- [Derived] Iglesia CB, Sokol AI, Sokol ER, Kudish BI, Gutman RE, Peterson JL, Shott S. Vaginal mesh for prolapse: a randomized controlled trial. Obstet Gynecol. 2010 Aug;116(2 Pt 1):293-303. doi: 10.1097/AOG.0b013e3181e7d7f8. PMID 20664388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 3, 2007 to August 1, 2009, 238 women were identified as eligible and 65 randomized (32 to experimental group (mesh) and 33 to control group (non-mesh)).
  All patients completed 3 month followup. Study recruitment halted at median followup of 9.7 months due to pre-determined criteria of vaginal mesh exposure in 5/32 patients (15.6%) in the mesh arm.
Groups:
- Prolift Mesh: vaginal prolapse repair with anterior or total mesh
  synthetic monofilament polypropylene mesh: Vaginal prolapse repair with mesh
- Prolapse Repair Without Mesh: vaginal prolapse repair without mesh (native tissue repair)
Period: 3 Months
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
Started | 32 | 33 (One originally randomized to the vaginal mesh arm but did not receive mesh due to inadequate vaginal caliber)
Completed | 32 | 33
Not Completed | 0 | 0
Period: 12 Months
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0
Period: 36 Months
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
Started | 33 (One of these was in the vaginal mesh arm but did not receive mesh due to inadequate vaginal caliber. For the 3 year outcomes, she was placed in the intent to treat but this was managed differently in the primary manuscript at 3 months and 1 year.) | 32
Completed | 25 | 26
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 1 | 2
Not completed — Censored due to reoperation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.6) | 63.1 (9) | 62.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 17 | 33
  African American | 6 | 7 | 13
  Hispanic | 2 | 2 | 4
  Asian | 1 | 0 | 1
Postmenopausal [Count of Participants; unit: Participants] | 23 | 24 | 47
Parity [Median (Inter-Quartile Range); unit: number deliveries] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (5.5) | 28.2 (6.4) | 27.9 (6.0)
POP-Q stage [Count of Participants; unit: Participants] — Stages of POP-Q system measurement:
  Stage 0 no prolapse is demonstrated
  Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen
  Stage 2 the most distal portion of the prolapse is 1 cm or less proximal or distal to the hymenal plane
  Stage 3 the most distal portion of the prolapse protrudes more than 1 cm below the hymen but protrudes no farther than 2 cm less than the total vaginal length (for example., not all of the vagina has prolapsed)
  Stage 4 vaginal eversion is essentially complete
  Participants
    stage 2 | 7 | 4 | 11
    stage 3 | 16 | 18 | 34
    stage 4 | 2 | 4 | 6
married [Count of Participants; unit: Participants] | 16 | 19 | 35
education [Count of Participants; unit: Participants]
  High school or less | 0 | 1 | 1
  completed high school | 4 | 8 | 12
  college or graduate | 21 | 17 | 38
insurance [Count of Participants; unit: Participants]
  Private | 12 | 12 | 24
  medicare | 13 | 14 | 27
hysterectomy [Count of Participants; unit: Participants] | 9 | 9 | 18
prior prolapse surgery [Count of Participants; unit: Participants] | 2 | 0 | 2
prior incontinence surgery [Count of Participants; unit: Participants] | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anatomic Cure at 3 Years
Description: 3 different measures for Anatomic cure using POPQ measurements:
  1. POP-Q at Stage I or less* (POP-Q points Ba, Bp or C -1 or less);
  2. no prolapse beyond the hymen (Ba, Bp or C 0 or less);
  3. no prolapse beyond the hymen (Ba, Bp 0 or less) with adequate apical support above the midvagina (C to TVL/2 or less) No bulge symptoms using Pelvic Floor Distress Inventory, PFDI question 3; do you see or feel a bulge in the vaginal area with response of no.
  Patient Satisfaction using Patient Global Impression of Improvement with response of very much better or much better
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
Number analyzed (Participants) | 25 | 26
Participants
  no reoperation/retreatment | 20 | 21
  composite stage less than/equal 1, no bulge symptoms, satisfaction very much better or much better | 8 | 8
  composite no prolapse beyond hymen, no bulge symptoms, satisfaction very much better or much better | 15 | 12
Statistical Analysis 1: Comparison: Prolift Mesh vs Prolapse Repair Without Mesh; Sample size primary outcome 1 year: 45 participants per arm, 20% difference success (70% no mesh and 90% mesh), alpha of .05 and 80% power, 15% loss to follow-up; Test type: Superiority — Statistical analysis was performed using SAS 9.1 software. One patient did not receive the assigned mesh treatment because the surgeon felt there was inadequate vaginal caliber, so non mesh repair was performed. This subject was analyzed in the non mesh group for the 3-month and 1-year outcomes rather than intent-to-treat approach. This subject was lost to follow-up after 12 months and not included in the 3-year analysis; p < 0.05, t-test, 2 sided; t-tests, Wilcoxon signed rank, Wilcoxon rank-sum tests continuous variables; X2 for categorical variables. Combined cure outcomes Fisher's exact test

2. Secondary Outcome: Bothersome Dyspareunia
Description: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire question 5 response of usually or always and tracked resolution, persistence, de novo dyspareunia
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
Number analyzed (Participants) | 14 | 11
Participants
  Persistent dyspareunia | 5 | 5
  resolution dyspareunia | 2 | 1
  de novo dyspareunia | 2 | 1

ADVERSE EVENTS:
Time Frame: 3 months, 1 year, 3 years
Arm/Group | Prolift Mesh | Prolapse Repair Without Mesh
All-Cause Mortality (participants affected / at risk) | 1/32 | 2/33
Serious Adverse Events (participants affected / at risk) | 5/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolift Mesh (N=32) | Prolapse Repair Without Mesh (N=33)
Surgery/reoperation for mesh exposure (Surgical and medical procedures) | 5 (5) | 0 (0) — Reoperation for mesh related complication, exposure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolift Mesh (N=32) | Prolapse Repair Without Mesh (N=33)
suture exposure (Surgical and medical procedures) | 0 (0) | 5 (5) — Gore-tex suture exposure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No